CLINICAL TRIAL: NCT00996242
Title: An Exploratory Open Label Study of Adjunctive L-lysine Treatment in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Birgitta Rembeck, PhD, The Sahlgrenska University Hospital, Gothenburg, Sweden
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LYSINE1; 07TGS-1049
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; L-lysine; PANSS
MeSH Terms: conditions — Schizophrenia | interventions — Lysine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- L-lysine (Experimental)
  Interventions: Drug: L-lysine

INTERVENTIONS:
Drug: L-lysine — 6 g/day for four weeks

SUMMARY:
The objective of the present study was to investigate the possibility of using L-lysine, an amino acid that occurs naturally in food and which interferes with nitric oxide (NO) production, for the treatment of schizophrenia. L-lysine, 6 g/day, was administered to ten patients with schizophrenia as an add-on treatment to conventional antipsychotic treatment. The study was designed as a single-blinded, cross-over study where patients were randomly assigned to initial treatment with either L-lysine or placebo and screened at baseline, after four weeks when treatment was crossed over, and after eight weeks when treatment was terminated. The four-week L-lysine treatment regimen caused a significant increased in blood concentration of the amino acid and was tolerated well. The analysis of outcome measures showed a significant decrease in symptom severity as measured by the Positive and Negative Syndrome Scale (PANSS). Furthermore, the patient's ability to solve the Wisconsin Card Sorting Task (WCST) was significantly improved indicating increased problem solving capacity and cognitive flexibility. Subjective reports from three of the patients also indicated decreased symptom severity and enhanced cognitive functioning. In summary, these findings suggest potential beneficial effects of L-lysine treatment on symptom severity and cognitive deficits in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* a stable phase of illness
* a stable dose of antipsychotic medication
* no other major medical conditions or other psychiatric diagnosis
* normal admission laboratory tests and vital signs

Exclusion Criteria:

* substance abuse, apart from smoking

Ages: 23 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Psychotic symptoms severity | Eight weeks

SECONDARY OUTCOMES:
Treatment safety assessment | Eight weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska Univeristy Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Wass C, Klamer D, Katsarogiannis E, Palsson E, Svensson L, Fejgin K, Bogren IB, Engel JA, Rembeck B. L-lysine as adjunctive treatment in patients with schizophrenia: a single-blinded, randomized, cross-over pilot study. BMC Med. 2011 Apr 18;9:40. doi: 10.1186/1741-7015-9-40. PMID 21501494